CLINICAL TRIAL: NCT06593769
Title: Glycemic and Appetite Effects of a Pre-meal Whey-Protein Microgel (the GAP Study)
Brief Title: Glycemic and Appetite Effects of a Pre-meal Whey-Protein Microgel
Acronym: GAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 2401CLI
Record Dates: First submitted 2024-07-11; First posted 2024-09-19 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Glucose Metabolism; Appetite Regulation
Keywords: glucose; appetite; proteins

STUDY DESIGN:
Intervention Model Description: Participants who meet the eligibility criteria will be randomized in 1:1 allocation ratio to one of the sequences (i.e., randomization groups):
  * sequence 1 = whey-protein microgel (WPM) in Day 2-Day 5 (period 1) and placebo in Day 9-Day 12 (period 2)
  * sequence 2 = placebo in period 1 and WPM in period 2. Randomization will be carried out using Medidata Rave RTSM.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Randomization sequence 1 (Other): Whey-protein microgel (day 2 -5); placebo (water) (day 9 to day 12) Crossover design - all participants will undergo the same experimental conditions
  Interventions: Dietary Supplement: whey-protein microgel; Other: Placebo
- Randomization sequence 2 (Other): Placebo (water) (day 2 -5); whey-protein microgel (day 9 to day 12) Crossover design - all participants will undergo the same experimental conditions
  Interventions: Dietary Supplement: whey-protein microgel; Other: Placebo

INTERVENTIONS:
Dietary Supplement: whey-protein microgel — The product used in this study is a liquid 125 mL whey protein microgel (WPM) formulation that will be delivered in a ready-to-drink formulation. The WPM is dairy based and, aside from milk and lactose, no other allergens are present Whey proteins and caseinates are two major fractions of cow milk proteins.
Other: Placebo — Water (isovoloumous amount)

SUMMARY:
In this study, the investigators want to assess the effects of a short-term twice daily pre-meal consumption of a liquid whey-protein microgel formulation, when compared to placebo (i.e., water), on:

* post-prandial glucose
* appetite This is an open-label study in 18 overweight or obese participants. This study will be performed in one center, the Clinical Innovation Laboratory (CIL), Nestlé Research, Lausanne. Participants will be screened and randomly assigned to 1 of 2 sequences of consumption. Enrolled participants will then consume the test product, or placebo, pre-breakfast and pre-lunch for four days and then crossover to the other product, over a period of 12 days.

DETAILED DESCRIPTION:
This study aims to provide new insights, and confirm a number of previous observations related to the role of whey-protein microgel in supporting glycemic regulation and supporting appetite regulation in people with overweight or obesity.

- Primary objective: The primary objective is to assess the effect of a pre-meal intake of whey-protein microgel (WPM) versus placebo on post-prandial glucose (PPG) response after a standardized breakfast meal in participants with BMI of 27 - 35 kg/m2, aged between 45 and 70 years.

Primary endpoint:

The primary endpoint is the 2-hour iAUC postprandial glucose (PPG) excursion induced by a standardized breakfast with pre-breakfast (-15 min) WPM compared to placebo.

- Secondary objectives: The secondary exploratory objective is to compare the effect of pre-meal (-15 min) intake (at breakfast and lunch) of WPM versus placebo on appetite and further glycemic parameters in participants with BMI of 27 - 35 kg/m2, aged between 45 and 70 years.

Secondary endpoints:

1. Hunger/fullness visual analogue scale scores and composite appetite scores onwards from pre-meal consumption of WPM or placebo (-15 min) during breakfast and lunch on visit days
2. Amount of food consumed during ad libitum lunch meal on visit days
3. 2-hour iAUC-15-120min of PPG excursion induced by an ad libitum lunch with pre-lunch (-15 min) WPM vs placebo
4. Mean 24h glucose from continuous glucose monitor (CGM) (Mean of day 2 (08:00 AM) to day 5 (08:00 AM) with placebo) vs Day 2-5 with WPM (same time period as without WPM)
5. Mean glucose from CGM considering only assumed "breakfast and lunch time measures" (08:00 AM - 04:00 PM) on day 2 - 4 between WPM and placebo
6. Glucose stability from CGM (mean 24h interquartile glucose range of day 2 (08:00 AM) to day 5 (08:00 AM) with placebo vs Day 2-5 with WPM (same time period as without product WPM)
7. Glucose stability from CGM considering only assumed "breakfast and lunch time measures" (mean interquartile glucose range of day 2-4 (08:00 AM - 04:00 PM) with placebo vs Day 2-4 with WPM (same time period as without product WPM)
8. Effects on primary and secondary exploratory endpoints by subgroups defined by median BMI

   The overall study implementation phase is expected to last for approximately 10 weeks. Expected duration of recruitment and screening procedures: up to 4 weeks. For logistical reasons, the participants will be divided in 2 groups with each group's study visits (V1 to V4) lasting 3 weeks each. The study is planned from Q2 to Q4 2024. This study will be conducted in compliance with the protocol, the current version of the Declaration of Helsinki, the ICH-GCP, the HRA as well as other locally relevant legal and regulatory requirements.

   - Sample size calculations and randomization A total of 15 participants (completers) will be required to detect an effect size of 0.56, representing a reduction of 20% in incremental AUC over 2h following the standardized breakfast (iAUC-15-120min) between WPM and placebo, within-subject correlation of 0.8, and a power of 90% at the 2-sided 5% significance level. Assuming a roughly 20% drop-out rate, 18 participants are planned for enrollment.

   Participants who meet the eligibility criteria will be randomized in 1:1 allocation ratio to one of the sequences (i.e., intervention groups): sequence 1 = WPM in Day 2 - Day 5 (period 1) and placebo in Day 9 - Day 12 (period 2) or sequence 2 = placebo in period 1 and WPM in period 2. Randomization will be carried out using Medidata Rave RTSM.

   - Statistical analysis Baseline characteristics (anthropometric measurements and blood laboratory measurements) will be summarized for all participants in the ITT set. Descriptive statistics of the laboratory blood measurements at baseline will be used to characterize the participants in the study. A complete set of descriptive statistics (records, mean, standard deviation, median, Q1 and Q3) will be provided for all data collected in the study. Data and results will be illustrated with figures (line plots and boxplots).

   For the analysis of the primary endpoint, the glucose iAUC-15-120min (incremental area under the curve in the time interval -15 min-120 minutes) will be extracted from the continuous glucose monitoring device at specific time points (15 minutes pre-breakfast, beginning of breakfast and then every 15 minutes after beginning of breakfast for 2 hours) on visit days V2, V3 and V4 respectively. For the comparison between WPM and placebo, a mixed linear model with response the glucose iAUC-15-120min will be proposed with fixed covariates: baseline blood glucose levels, treatment, and period (period 1 or period 2). Participant identifier will be used as random effect. For this efficacy study, the FAS dataset is the population of primary interest to conclude on the primary objective with support from the per protocol dataset. As an exploratory model for the analysis of the primary endpoint, the curves of the continuous glucose monitoring in the time interval 15 minutes pre-breakfast to 2 hours after the beginning of breakfast on days V2, V3 and V4 respectively will be the responses of a functional mixed linear model with the same covariate as the linear mixed model explained above (baseline blood glucose levels, treatment arm and period).

   For the Hunger/Fullness VAS score calculation, the iAUC will be estimated as the sum of the areas located above the baseline value

   - Datasets to be analysed Intention-to-treat (ITT) analysis population: all randomized participants. Safety analysis set (SAF) analysis population: safety data (e.g., adverse events) are analyzed in the SAF which consists of all participants in the ITT population with documentation of at least one administration of study product, i.e. whey protein microgel or placebo.

   Full Analysis Set (FAS) analysis population: the FAS dataset includes all participants/infants from SAF (participants that took at least one dose of study product or placebo) without participants who failed to satisfy study entry eligibility criteria or had no post-randomization data.

   Per Protocol (PP) analysis population: PP dataset consists of participants/infants from the FAS without any departures from the protocol which are believed to impact the primary analysis.

   - Study Monitoring The monitoring will be performed by the Centre de recherche Clinique (CRC) at CHUV (Lausanne). Monitoring visits allow the sponsor representative to evaluate study progress, verify accuracy and completeness of eCRFs, resolve any inconsistencies in the study records, and ensure that all protocol requirements, applicable local laws, ICH guidelines, and investigator obligations are fulfilled. The monitoring activities will be performed at agreed times during the study and after the study has been completed. The extent, schedule, and nature of monitoring activities based on the objective and design of the study are defined in a study specific monitoring plan, drafted by the Clinical Project Manager (CPM) from the sponsor side, and agreed upon and signed by the representatives of the external monitor, the sponsor CPM, and the sponsor Clinical Data Manager. The investigator will allow sponsor representatives to periodically review the eCRF and corresponding office, hospital, and laboratory records (source documents) of each study participant. Case report forms must be completed by the Investigator on a regular basis and prior to each monitoring visit.
   * Data sources Most of data will be entered from the source document into an electronic Case Report Forms (eCRF - web database) entitled RAVE, solution of iMedidata. For some questionnaires, data will be entered directly by the participant in an ePRO Medidata, as source data transmitted automatically into the eCRF. Data should be entered in eCRF within 7 days after the participant's visit. At the end of the study, the Principal Investigator must sign each eCRF electronically.

   Investigator's site data: site personnel will directly enter these data into the eCRF via manual data entry. The exhaustive list of data collected at each visit will be described in the Data Listing document. The Data Listing document is written by the Clinical Data Manager (CDM) and approved by the Clinical Team. All the site source documents are listed in the Source Data Log available in the related investigator file.

   Participant reported outcome: the following questionnaires/diaries will be considered as Source document and entered by participant in ePRO. The ePRO is directly linked to the eCRF and these data are automatically captured in the eCRF:

   • The "Hunger/Fullness VAS Questionnaire" will be considered as a source document and entered by the participant at site on scheduled time points on paper. Records will be measured and entered into the eCRF by the study site staff.

   • The "Product Intake Compliance Questionnaire" ePRO notebook will be considered as a source document and entered by the participant at home on scheduled timepoints. Records will be verified in the eCRF by the study site staff.

   • The "Adverse Events and Concomitant Medications Diary" ePRO notebook will be considered as a source document and entered by the participant at home available at any time. Records will be verified in the eCRF by the study site staff and additional information clarified.

   External clinical and laboratory data: in addition to the data recorded in the eCRF, the laboratory results will be entered into Labkey database to be transferred into Life Science Analytics Framework (LSAF) for analysis and storage.

   The CGM data will be extracted through a local software and collected at site during the study visits. The raw data files will be reconciled by CDM and stored in LSAF for further data analysis. To ensure traceability, the files will be downloaded in CSV format and converted into PDF. Once converted, each PDF file will be entitled using the participant ID and the visit date, dated and electronically signed by the investigator. The files will be then archived in Investigator Site Files.

   - Data Validation The CDM will validate all data entered into the eCRF. All computerized edit checks programmed to validate the data, at least on primary data outcome, are described in the Data Validation Plan document, written by the CDM.

   Data discrepancies will trigger automatic queries, directly displayed on the screen when data entered are saved. Manual Data Reports will be produced by CDM for review by the team regularly. If necessary, manual queries will be sent to the Investigator for clarification. All these discrepancies/queries must be documented, answered, or confirmed by the site using Medidata Query tools.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females aged 45 - 70 years, at enrolment.
2. Body mass index (BMI) ≥ 27 kg/m² but < 35 kg/m².
3. Healthy participants based on medical history.
4. Able to understand and to sign a written informed consent prior to study enrolment.
5. Willing and able to comply with the requirements for participation in this study.

Exclusion Criteria:

1. Any past or on-going diagnosed medical/surgical condition (i.e., diabetes, malignancy, gastrointestinal disease, chronic inflammatory condition, chronic kidney disease, cardiovascular disease, bleeding disorder) and/ or psychiatric condition (e.g. depression, psychotic disorders, chronic insomnia, eating disorder), which in the opinion of the site physician/investigator may risk participant's well-being/safety, impede participant compliance with study procedures or ability to complete the study and/or could confound the primary objectives of the study.
2. Random plasma glucose ≥ 11.1 mmol/L or fasting plasma glucose ≥ 7.0 mmol/L (finger-prick point-of-care [POC] testing)
3. HbA1c ≥ 6.5% (finger-prick POC testing)
4. Known inborn errors of amino acid and protein metabolism.
5. With planned/scheduled medical imaging procedure/s (magnetic resonance imaging [MRI], computed tomography [CT] scan, X-ray), or electrical heat (diathermy) treatment during the study period.
6. Known or suspected allergies or intolerances to any of the ingredients of the nutritional formulation (i.e., milk, lactose) and the study meals.
7. Known or suspected cutaneous hypersensitivity to adhesives, silicon, or plaster.
8. Substantial changes in eating habits (i.e., switching from one dietary regimen to another) up to 30 days before enrolment.
9. Anticipated change in usual physical activity levels during the study period (e.g., plans for undertaking new vigorous-intensity physical activity such as: jogging, running, carrying heavy objects or other loads upstairs, shoveling snow, participating in a fitness class, and fast swimming, that will lead to hard and fast breathing).
10. Any chronic alcohol or drug abuse within the past year; specifically, alcohol intake > 2 servings per day for males and >1 serving per day for females. A serving corresponds to 0.35dl of liquor/strong alcohol, 1 dl of wine, or 3 dl of beer.
11. Female participants who are pregnant, lactating and/or breastfeeding.
12. Participants who refuse to be informed of incidental findings relevant to their health (e.g. abnormal laboratory results).
13. Currently participating in another interventional study.
14. Family or hierarchical relationships with the research team members.

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2024-10-09 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2024-12-23 (Actual)

PRIMARY OUTCOMES:
Post-prandial glucose - by continuos glucose measurement software | V2 (day 1), V3 (day 5), V4 (day 12)
  The effect of a pre-meal intake of WPM versus placebo on PPG response after a standardized meal in participants with BMI of 27 - 35 kg/m2.

SECONDARY OUTCOMES:
Appetite regulation - through a VAS questionnaire | V2 (day 1), V3 (day 5), V4 (day 12)
  Hunger/fullness visual analogue scale (VAS) scores onwards from pre-meal consumption of WPM or placebo (-15 min) during breakfast (1h-, 2h-, and 3h-iAUC) and lunch (1h-, and 2h-iAUC) on visit days
Appetite regulation - composite score - through a VAS questionnaire | V2 (day 1), V3 (day 5), V4 (day 12)
  Composite appetite score (CAS) onwards from pre-meal consumption of WPM or placebo (-15 min) during breakfast (1h-, 2h-, and 3h-iAUC) and lunch (1h-, and 2h-iAUC) on visit days
Ad libitum food intake - weighted on the scale | V2 (day 1), V3 (day 5), V4 (day 12)
  Amount of food consumed during ad libitum lunch meal on visit days
Effect of the intervention on the post-prandial glucose after an ad libitum lunch | V2 (day 1), V3 (day 5), V4 (day 12)
  2-hour iAUC-15-120min of PPG excursion induced by an ad libitum lunch with pre-lunch (-15 min) WPM vs placebo
Mean daily glucose, intervention vs placebo - by continuos glucose measurement software | Day 2 (08:00 AM) to day 5 (08:00 AM) (3 days in total)
  Mean 24h glucose from continuous glucose monitor (CGM), WPM vs placebo (water)
Glucose stability, intervention vs placebo - by continuos glucose measurement software | Day 2 (08:00 AM) to day 5 (08:00 AM) (3 days in total)
  Mean 24h interquartile glucose range from CGM, WPM vs placebo (water)
Glucose stability, intervention vs placebo, only breakfast/lunch - by continuos glucose measurement software | Day 2 (08:00 AM) to day 5 (08:00 AM) (3 days in total)
  Mean interquartile glucose range from CGM considering only assumed "breakfast and lunch time measures"
Anthropometric measurements: weight - through a scale | V2 (day 1)
  Median weight (in kg)
Anthropometric measurements: height - through a scale | V2 (day 1)
  Median height (in mt)
Subgroup analysis by Body Mass Index (BMI) (kg/m^2) | Through the study, from V2 until V4 (12 days in total)
  Effects on primary and secondary exploratory endpoints by subgroups defined by median BMI. Weight and height will be combined to report BMI in kg/m^2 as it follows: BMI (kg/m^2) = weight (kg) / height^2 (m^2)

CONTACTS AND LOCATIONS:
Overall Officials: Nora Schneider, Principal Investigator — Nestlé Research
Locations (1):
- Clinical Innovation Laboratory, Lausanne, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Neeland IJ, Tsintzas K, Ahren B, Chilton RJ, Giorgetti A, Mondragon A, Ambiaux R, Migliavacca E, Philippe D, Aprikian O, Johansen OE. Short-term pre-meal whey protein microgel supplementation reduces postprandial glycemia and appetite in adults with overweight: An open-label randomised controlled trial. Obes Pillars. 2025 May 26;15:100183. doi: 10.1016/j.obpill.2025.100183. eCollection 2025 Sep. PMID 40521305